CLINICAL TRIAL: NCT02626949
Title: Effects of Mindfulness Training on Chronic Inflammation in HIV-Infected Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jeffrey J Weiss, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 13-1990; 1R21AT008540-01 (NIH)
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: HIV
Keywords: HIV; AIDS; Mindfulness; Mindfulness-based stress reduction; Stress; Intervention; Inflammation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Inflammation | interventions — Mindfulness; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MBSR Course (Experimental): Mindfulness-Based Stress Reduction Course (MBSR) consisting of 8 weekly sessions, 2.5 hours each, and a 5 hour silent retreat during the 6th week of the program.
  Interventions: Behavioral: MBSR Course
- HEP Course (Experimental): Health Enhancement Program (HEP) consisting of 8 weekly sessions, 2.5 hours each, and 1.5 hour monthly educational sessions after the 8 week intervention.
  Interventions: Behavioral: HEP Course

INTERVENTIONS:
Behavioral: MBSR Course — Formal mindfulness meditation methods taught in the MBSR course include: Body Scan Meditation (a supine meditation), Gentle Hatha Yoga (practiced with mindful awareness of the body), Sitting Meditation (mindfulness of breath, body, feelings, thoughts, and emotions), and Walking Meditation. Informal Mindfulness Meditation Practices (mindfulness in everyday life) include: 1) awareness of pleasant and unpleasant events, and, 2) deliberate awareness of routine activities and events such as eating, weather, walking, and interpersonal communication. Daily home assignments include a minimum of 30 minutes daily formal mindfulness practices and 5-15 minutes informal practice, 6 days per week for the entire duration of the course. Course sessions will consist of discussions oriented around weekly homework assignments, including an exploration of obstacles, and development of self-regulatory skills and capacities.
  Other Names: Mindfulness meditation; Mindfulness-Based Stress Reduction
  Arms: MBSR Course
Behavioral: HEP Course — HEP is an active control that matches MBSR in non-specific factors, such as the amount of time participants interact, but does not include mindfulness practice as an active component. HEP instructors will be selected from experts in the areas covered: music, nutrition education, and, functional movement. The study's RC will coordinate HEP sessions and monitor attendance. Following the 8-week HEP protocol, subjects will meet monthly in 1.5-hour educational sessions to match the booster sessions of MBSR participants.
  Other Names: Health Enhancement Program
  Arms: HEP Course

SUMMARY:
By 2015 half of the people living with HIV infection in the U.S. are estimated be over the age of 50, and this cohort of patients with well-controlled plasma viremia is aging at a more rapid pace than their non-HIV peers. Long-term chronic inflammation plays a critical role in premature aging in HIV-infected adults. Markers associated with chronic inflammation, including IL-6, CRP, sCD14 and d-dimer, have not only been shown to be present at higher levels in HIV-infected adults, but are also correlated to a wide variety of morbidities and mortality. The goal of this project is to determine the impact of two different interventions -- Mindfulness-Based Stress Reduction (MBSR) and Health Enhancement Program (HEP) -- on reducing biological markers associated with chronic inflammation in HIV-infected adults with an undetectable HIV viral load. In order to achieve this goal, a pilot RCT with 120 subjects over 50 years old who are on anti-retroviral therapy (ART) will be conducted with the following specific aims: 1) to assess the effect of MBSR and/or HEP on biomarkers of chronic inflammation (IL-6, CRP, sCD14, d-dimer), and, 2) to explore whether changes in psychological well-being (anxiety, depression, fatigue, cognitive functioning) mediate the impact on chronic inflammation. Subjects will be randomized to participation in a group MBSR course or to the HEP group both of which consist of 8 weekly sessions followed by 6 monthly booster sessions. Three time points will be measured: baseline, 8 weeks (immediately after completion of weekly intervention), and 6-months post-completion of weekly intervention. Mixed linear and structural equation model will be used to test the study hypotheses. The proposed study is innovative in that it is the first to explore the impact of a complementary mind-body intervention on chronic inflammation in HIV-infected adults. Given that the consequences of early aging in this cohort will be a burden on the health care system as well as a medical, social and psychological burden on those living with HIV, the study has the potential to have a major public health impact.

DETAILED DESCRIPTION:
The proposed study will be the first to examine any form of alternative or complementary holistic therapy in older long-term HIV-infected persons with well-controlled plasma viremia. It will also be the first mind-body study of HIV-infected adults to be conducted using the most rigorous randomized controlled trial (RCT) design. From a translational medicine perspective, this study is innovative in that it examines a comprehensive set of biological markers specifically associated with chronic inflammation. No previous mind-body study has specifically targeted a set of biological markers that not only have been proven to be elevated in adults with HIV, but also been described as predictors of morbidity and overall mortality. This would be the first study to explore whether improvements in markers of psychosocial stress mediate the impact of the proposed interventions on chronic inflammation.

This study is innovative in its effort to move HIV care beyond the current focus on virologic control, optimization of comorbid conditions, and encouragement of healthy lifestyle to include active interventions that can address the state of chronic inflammation and immune dysfunction underlying the early and accelerated aging process. Most bio-behavioral research in HIV to date has understandably focused on patients with poor adherence to HIV medication and treatment. This study is novel in its focus on highly adherent patients and the significant changes in profiles of biological markers associated with chronic inflammation documented in this cohort. The complementary medicine approach being studied has the potential to be integrated into the existing healthcare paradigm for HIV-positive persons.

Specific Aims:

Aim 1: To assess the effect of MBSR and HEP on biomarkers of chronic inflammation (IL-6, CRP, sCD14, d-dimer), in HIV-infected adults with well-controlled plasma viremia.

Aim 2: To explore whether changes in markers of psychosocial well-being (anxiety, depression, fatigue, cognitive functioning) mediate the impact of these mind-body interventions on chronic inflammation.

General Study Design: The proposed study is a prospective, randomized, clinical trial with attention control under the direction of the dual PIs, a behavioral scientist and a virologist. The study team is also made up of investigators from infectious diseases, mind-body medicine, geriatrics, and biostatistics. Subjects will be randomized to participation in an 8-week group MBSR course or to the Health Enhancement Program (HEP). The study population will consist of 120 individuals, 50 years old or older, long-term (5 years on ART or longer) HIV-infected adults with well-controlled plasma viremia and baseline IL-6 level of 1.17 pg/mL or greater. Randomization will be stratified to achieve balanced distribution between the groups based on gender and study site. One cohort group will participate in the 8-week MBSR course followed by six, once-per-month booster sessions, and separate cohort group will participate in HEP, with additional monthly educational meetings for six months. Both groups will be evaluated using two sets of measures: biological markers associated with chronic inflammation (IL-6, CRP, sCD14, d-dimer) and measures of psychosocial stress (anxiety, depression, fatigue, and mindfulness). Subjects will be assessed at three time points: baseline, 8 weeks (immediately after completion of weekly interventions), and 6-months post weekly courses (immediately after completion of booster sessions). The investigators will use mixed linear and structural equation model to test study hypotheses.

ELIGIBILITY:
Inclusion criteria:

* HIV-infected for 5 or more years
* On ART for 5 or more years
* HIV viral load consistently <48 copies/mL for the last year
* No anticipated changes in ART by provider or patient
* Fluency in the English language
* Age 45 years or older
* Willingness to complete the entire MBSR or HEP interventions

Exclusion criteria:

* Having participated in an MBSR course in the past
* Current meditation and/or yoga practice
* Began psychiatric medications in the past 2 months or plans to discontinue psychiatric medications
* Currently receiving steroids or immunosuppressant drugs
* Women who are pregnant or plan to become pregnant in the next year

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weiss, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Peter Barbosa, PhD, Principal Investigator — New York College of Podiatric Medicine
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 114 were randomized prior to enrollment with final participants enrollment of 84.
Groups:
- MBSR Course: Mindfulness-Based Stress Reduction Course (MBSR) consisting of 8 weekly sessions, 2 hours each, and a 5 hour silent retreat during the 6th week of the program.
- HAEP Course: Health & Arts Enrichment Program (HAEP) consisting of 8 weekly sessions, 2 hours each, and 5 hour educational session during the 6th week of the program.
Period: Randomization, Pre-Enrollment
Arm/Group | MBSR Course | HAEP Course
Started | 56 | 58
Completed | 40 | 44
Not Completed | 16 | 14
Not completed — did not attend the baseline interview | 15 | 11
Not completed — did not meet inclusion criteria post-randomization | 1 | 3
Period: Enrolled
Arm/Group | MBSR Course | HAEP Course
Started | 40 | 44
Completed | 30 | 36
Not Completed | 10 | 8
Not completed — Lost to Follow-up | 7 | 6
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MBSR Course | HAEP Course | Total
Number analyzed (Participants) | 40 | 44 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (5.9) | 59.0 (7.4) | 58.3 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 21 | 26 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 15 | 31
  Not Hispanic or Latino | 24 | 29 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 26 | 52
  White | 14 | 18 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Interleukin 6 (IL-6) Biological Markers
Description: Interleukin 6 (IL-6) biological markers at 8 weeks and 6 months as compared to baseline.
Time Frame: Baseline, 8 weeks post intervention, and 6 months post intervention
Population: One participant did not have data for baseline. Data for those participants who completed the 8 weeks and 6 months post-intervention included.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | MBSR Course | HAEP Course
Number analyzed (Participants) | 40 | 44
pg/mL
  Baseline: number analyzed (Participants) | 39 | 44
  Baseline | 2.24 [1.48 to 3.69] | 2.63 [1.41 to 3.70]
  8 weeks (post intervention): number analyzed (Participants) | 33 | 40
  8 weeks (post intervention) | 2.53 [1.73 to 4.34] | 2.88 [1.59 to 3.75]
  6 months (post intervention): number analyzed (Participants) | 30 | 37
  6 months (post intervention) | 2.89 [1.61 to 5.69] | 2.62 [1.39 to 4.91]

2. Secondary Outcome: PROMIS - Anxiety
Description: Patient Reported Outcomes Measurement Information System (PROMIS) - Anxiety - Measures of Psychosocial Stress, total scale 5-40 with higher score indicating more anxiety
Time Frame: Baseline, 8 weeks post intervention, and 6 months post intervention
Population: Data for those participants who completed the 8 weeks and 6 months post-intervention included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBSR Course | HAEP Course
Number analyzed (Participants) | 40 | 44
score on a scale
  Baseline | 18.7 (8.2) | 19.3 (6.9)
  8 weeks post intervention: number analyzed (Participants) | 33 | 39
  8 weeks post intervention | 15.1 (6.6) | 18.4 (7.4)
  6 months post intervention: number analyzed (Participants) | 30 | 36
  6 months post intervention | 15.9 (6.9) | 18.5 (7.5)

3. Secondary Outcome: PROMIS - Fatigue
Description: Patient Reported Outcomes Measurement Information System (PROMIS) - Fatigue - Measures of Psychosocial Stress, total scale 5-40 with higher score indicating more fatigue
Time Frame: Baseline, 8 weeks post intervention, and 6 months post intervention
Population: Data for those participants who completed the 8 weeks and 6 months post-intervention included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBSR Course | HAEP Course
Number analyzed (Participants) | 40 | 44
score on a scale
  Baseline | 21.2 (8.1) | 21.4 (9.4)
  8 weeks post intervention: number analyzed (Participants) | 33 | 39
  8 weeks post intervention | 16.8 (7.7) | 21.1 (8.1)
  6 months post intervention: number analyzed (Participants) | 30 | 36
  6 months post intervention | 18.8 (8.0) | 19.3 (9.6)

4. Secondary Outcome: BDI-II
Description: Beck Depression Inventory (BDI-II) - Measures of Psychosocial Stress, total scale from 0-63, with higher score indicating more depression
Time Frame: Baseline, 8 weeks post intervention, and 6 months post intervention
Population: Data for those participants who completed the 8 weeks and 6 months post-intervention included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBSR Course | HAEP Course
Number analyzed (Participants) | 40 | 44
score on a scale
  Baseline | 15.0 (10.0) | 15.6 (10.6)
  8 weeks post intervention: number analyzed (Participants) | 33 | 39
  8 weeks post intervention | 9.7 (9.8) | 14.7 (10.6)
  6 months post intervention: number analyzed (Participants) | 30 | 36
  6 months post intervention | 9.7 (7.8) | 13.1 (11.7)

5. Secondary Outcome: FFMQ
Description: The Five Facet Mindfulness Questionnaire (FFMQ) - Measures of Mindfulness, full scale from 39 - 195, with higher score indicating more mindfulness
Time Frame: Baseline, 8 weeks post intervention, and 6 months post intervention
Population: Data for those participants who completed the 8 weeks and 6 months post-intervention included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBSR Course | HAEP Course
Number analyzed (Participants) | 40 | 44
score on a scale
  Baseline | 135.7 (21.8) | 135.4 (19.8)
  8 weeks post intervention: number analyzed (Participants) | 33 | 39
  8 weeks post intervention | 144.3 (18.6) | 134.7 (22.3)
  6 months post intervention: number analyzed (Participants) | 30 | 36
  6 months post intervention | 145.3 (19.2) | 141.5 (23.0)

6. Secondary Outcome: Retention Rates
Description: Attendance records will provide retention rates.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | MBSR Course | HAEP Course
Number analyzed (Participants) | 40 | 44
Participants | 30 | 36

ADVERSE EVENTS:
Time Frame: Adverse events collected from baseline to 8 weeks post-intervention
Arm/Group | MBSR Course | HAEP Course
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/44
Other Adverse Events (participants affected / at risk) | 0/40 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT02626949/Prot_SAP_000.pdf